CLINICAL TRIAL: NCT04989686
Title: Microsampling Assays for Immunosuppressive Drugs in Children
Acronym: MAIDEN
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-020410; 5R21HD106103-02 (NIH)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Immunosuppression
Keywords: microsampling; cyclosporine A; tacrolimus; sirolimus; Tasso-M20

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Investigators will plan to enroll up to 150 subjects to obtain 120 evaluable subjects (CYA: 40 subjects, SIR: 40 subjects, and TAC: 40 subjects).
  Two blood samples for up to five blood tests will be drawn simultaneously.
  1. Sample Collection 1 will be obtained from venous or arterial blood.
     1. Blood test 1: TDM measure of the immunosuppressive drug
     2. Blood test 2: Hemoglobin/hematocrit measurement (if not obtained as the standard of care within 12 hours prior or simultaneous with TDM measure will be obtained as a research collection)
  2. Sample collection 2 will be obtained from capillary blood through the Tasso-M20 device a. Blood test 3: Research indicated measurement of immunosuppressive drug concentration.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cyclosporine A: 1. Males and females <18 years of age
  2. Weight greater than 5 kg
  3. Receiving cyclosporine A as the standard of care
  4. Has scheduled/anticipated blood draw to quantify the concentration of cyclosporine A for clinical indications
  5. Parental/guardian permission (informed consent), and subject's assent if applicable.
  Interventions: Other: Microsampling
- Tacrolimus: 1. Males and females <18 years of age
  2. Weight greater than 5 kg
  3. Receiving tacrolimus as the standard of care
  4. Has scheduled/anticipated blood draw to quantify the concentration of tacrolimus for clinical indications
  5. Parental/guardian permission (informed consent), and subject's assent if applicable.
  Interventions: Other: Microsampling
- Sirolimus: 1. Males and females <18 years of age
  2. Weight greater than 5 kg
  3. Receiving sirolimus as the standard of care
  4. Has scheduled/anticipated blood draw to quantify the concentration of sirolimus for clinical indications
  5. Parental/guardian permission (informed consent), and subject's assent if applicable.
  Interventions: Other: Microsampling

INTERVENTIONS:
Other: Microsampling — Volumetric absorptive microsampling (VAMS) with Tasso-M20 devices allows for the accurate and precise collection of a fixed small volume of blood from a capillary needle without the need for phlebotomy.

SUMMARY:
Immunosuppressive therapy is used to treat and manage solid organ and bone marrow/stem cell transplants in children. However, it can be harmful if too little or too much is given. Monitoring immunosuppressive drug (cyclosporine A, tacrolimus, and sirolimus) concentrations in the blood is important to ensure that the drug is given safely and effectively, but current approaches for collecting blood from a vein are painful and often difficult in children. Investigators seek to compare a new approach for monitoring immunosuppressive drug concentrations using a novel small volume blood sampling device, called Tasso-M20, to the traditional way of collecting blood from a vein. Additionally Investigators are interested in assessing patient and family perceptions of the Tasso-M20 device being used for immunosuppressive therapy and their comfortability using the device outside of a clinical setting.

The primary objective of this project is to identify the relationship between cyclosporine A (CYA), tacrolimus (TAC), and sirolimus (SIR) concentrations in the venous blood (gold-standard) and capillary whole blood obtained using the microsampling device Tasso-M20.

The secondary objective of this study is to investigate the stability of CYA, TAC, and SIR in blood samples collected using the Tasso-M20 device under the conditions of shipping and storage.

The sub-study objective is to thematically compare subjects' and families' perceptions of blood collection via the Tasso-M20 device and standard venous blood collection.

DETAILED DESCRIPTION:
Immunosuppressive therapy is used to treat and manage solid organ and bone marrow/stem cell transplants; however, suboptimal dosing can lead to organ rejection and graft failure. Immunosuppressant drugs require therapeutic drug monitoring (TDM) to ensure dosing is adequate and therapeutic concentrations are achieved and maintained. The optimal blood concentrations of these drugs are critical to minimize toxicity and simultaneously prevent allograft rejection in an individual transplant patient. Often life-long TDM is required necessitating hospital or laboratory visits for routine venous blood sampling by phlebotomy. Immunosuppressive drugs, cyclosporine A (CYA), tacrolimus (TAC), and sirolimus (SIR) require routine TDM. This entails immunocompromised people leaving their homes for laboratory visits, potentially increasing their risk of acquiring infections.

TDM for CYA, TAC, and SIR are required due to their narrow therapeutic targets: CYA 150-400 ng/mL, TAC 5-12 ng/mL, and SIR 4-12 ng/mL. CYA, TAC, and SIR are primarily distributed in erythrocytes and should be quantified in whole blood. Immunoassays and the liquid chromatography-tandem mass spectrometry (LC-MS/MS) assays are the two commonly used methods of TDM for CYA, TAC, and SIR. While immunoassays provide an accurate measurement of concentrations, they often have some limitations on specificity. LC-MS/MS assays are very specific and efficient since they can quantify multiple analytes with a single method. At the Children's Hospital of Philadelphia (CHOP), the clinical TDM immunoassays for CYA, TAC, and SIR require 0.5-1.0 mL of blood. TDM immunoassays require blood collection by a trained practitioner.

Volumetric absorptive microsampling (VAMS) with an FDA-approved Tasso-M20 device allows for the accurate and precise collection of a fixed volume of blood from a capillary needle without the need for phlebotomy. The Tasso-M20 (FDA Class 1 exempt device) consists of a sample head with a lancet that is activated with the push of a button to accurately and painlessly collect blood samples from the deltoid (or similar) muscle (capillary sampling) of the subjects on all four tips (17.5 µL each). An LC-MS/MS assay with 20 µL blood, as obtained by the Tasso device, was shown to provide the required test range for TDM of trough values. This microsampling technique could be utilized clinically to promote the provision of TDM in children but has not been studied for immunosuppressive drugs (CYA, TAC, and SIR) in children.

Children and their parents/guardians who consent to the optional sub-study will be administered a brief survey after one study visit, to ask about their perceptions of the two methods of blood collection that they experienced at the visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females <18 years of age
2. Weight greater than 5 kg
3. Receiving CYA, TAC, and/or SIR as standard of care
4. Has scheduled/anticipated blood draw to quantify the concentration of CYA, TAC, and SIR* for clinical indications
5. Parental/guardian permission (informed consent), and subject's assent if applicable.

Exclusion Criteria:

1) Unable to provide blood samples.

* Potential subjects and their parents/guardians may be approached prior to having a blood draw scheduled if they meet all other eligibility criteria.

Sub-Study Criteria:

Sub-study criteria for child participants will not differ from the main study. Adult participants are required to be a parent/legal guardian of a study subject.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children receiving immunosuppressive therapy and scheduled/anticipated blood draw to quantify the concentration of the immunosuppressive drugs (CYA, TAC, and SIR) for clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical validation of microsampling assay of Tacrolimus | up to 20 months
  Capillary whole blood specimens will be obtained via the Tasso M-20 sampling device to determine validity of the assay compared to venous blood samples (gold standard and used clinically) in measuring Tacrolimus concentration levels.
Clinical validation of microsampling assay of Sirolimus | up to 20 months
  Capillary whole blood specimens will be obtained via the Tasso M-20 sampling device to determine validity of the assay compared to venous blood samples (gold standard and used clinically) in measuring Sirolimus concentration levels.
Clinical validation of microsampling assay of Cyclosporine A | up to 20 months
  Capillary whole blood specimens will be obtained via the Tasso M-20 sampling device to determine validity of the assay compared to venous blood samples (gold standard and used clinically) in measuring Cyclosporin A concentration levels.

SECONDARY OUTCOMES:
Stability of blood samples which contains immunosuppressive drug Tacrolimus under conditions of shipping | up to 20 months
  Blood specimens obtained by the Tasso M20 device will be used to investigate the stability of blood samples obtained from the Tasso M-20 device containing immunosuppressive drugs Tacrolimus under the conditions of shipping
Stability of blood samples obtained which contains immunosuppressive drug Sirolimus under conditions of shipping | up to 20 months
  Blood specimens obtained by the Tasso M20 device will be used to investigate the stability of blood samples obtained from the Tasso M-20 device containing immunosuppressive drugs sirolimus under the conditions of shipping
Stability of blood samples containing immunosuppressive drug Cyclosporine A under conditions of shipping | up to 20 months
  Blood specimens obtained by the Tasso M20 device will be used to investigate the stability of blood samples obtained by the Tasso M-20 device which contains immunosuppressive drugs cyclosporine A under the conditions of shipping
Stability of blood samples which contains immunosuppressive drug Tacrolimus under conditions of storage | up to 20 months
  Blood specimens obtained by the Tasso M20 device will be used to investigate the stability of blood samples containing immunosuppressive drugs Tacrolimus under the conditions of storage
Stability of blood samples which contains immunosuppressive drug Sirolimus under conditions of storage | up to 20 months
  Blood specimens obtained from the Tasso device will be used to investigate the stability of blood samples containing immunosuppressive drugs Sirolimus under the conditions of storage
Stability of blood samples obtained which contains immunosuppressive drug Cyclosporine A under conditions of storage | up to 20 months
  Blood specimens obtained from the Tasso M20 device will be used to investigate the stability of blood samples containing immunosuppressive drugs Cyclosporin A under the conditions of storage

OTHER OUTCOMES:
Usability of the two methods of blood collection | up to 20 months
  Usability will be measured by assessing participants survey responses about their perceptions of blood collection methods they experienced
Acceptability of the two methods of blood collection | up to 20 months
  Acceptability will be measured by assessing participants survey responses about their perceptions of blood collection methods they experienced

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Phildelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Enderby C, Keller CA. An overview of immunosuppression in solid organ transplantation. Am J Manag Care. 2015 Jan;21(1 Suppl):s12-23. PMID 25734416
- [Background] Penack O, Marchetti M, Ruutu T, Aljurf M, Bacigalupo A, Bonifazi F, Ciceri F, Cornelissen J, Malladi R, Duarte RF, Giebel S, Greinix H, Holler E, Lawitschka A, Mielke S, Mohty M, Arat M, Nagler A, Passweg J, Schoemans H, Socie G, Solano C, Vrhovac R, Zeiser R, Kroger N, Basak GW. Prophylaxis and management of graft versus host disease after stem-cell transplantation for haematological malignancies: updated consensus recommendations of the European Society for Blood and Marrow Transplantation. Lancet Haematol. 2020 Feb;7(2):e157-e167. doi: 10.1016/S2352-3026(19)30256-X. PMID 32004485
- [Background] Baert F, Vermeire S, Noman M, Van Assche G, D'Haens G, Rutgeerts P. Management of ulcerative colitis and Crohn's disease. Acta Clin Belg. 2004 Sep-Oct;59(5):304-14. doi: 10.1179/acb.2004.045. PMID 15641402
- [Background] Cheng-Lai A, Frishman WH. Sirolimus-eluting coronary stents: novel devices for the management of coronary artery disease. Am J Ther. 2004 May-Jun;11(3):218-28. doi: 10.1097/00045391-200405000-00011. PMID 15133538
- [Background] Zhang Y, Zhang R. Recent advances in analytical methods for the therapeutic drug monitoring of immunosuppressive drugs. Drug Test Anal. 2018 Jan;10(1):81-94. doi: 10.1002/dta.2290. Epub 2017 Sep 28. PMID 28851030
- [Background] Wallemacq P, Goffinet JS, O'Morchoe S, Rosiere T, Maine GT, Labalette M, Aimo G, Dickson D, Schmidt E, Schwinzer R, Schmid RW. Multi-site analytical evaluation of the Abbott ARCHITECT tacrolimus assay. Ther Drug Monit. 2009 Apr;31(2):198-204. doi: 10.1097/FTD.0b013e31819c6a37. PMID 19258928
- [Background] Veenhof H, Koster RA, Junier LAT, Berger SP, Bakker SJL, Touw DJ. Volumetric absorptive microsampling and dried blood spot microsampling vs. conventional venous sampling for tacrolimus trough concentration monitoring. Clin Chem Lab Med. 2020 Sep 25;58(10):1687-1695. doi: 10.1515/cclm-2019-1260. PMID 32412437
- [Background] Klak A, Pauwels S, Vermeersch P. Preanalytical considerations in therapeutic drug monitoring of immunosuppressants with dried blood spots. Diagnosis (Berl). 2019 Mar 26;6(1):57-68. doi: 10.1515/dx-2018-0034. PMID 30808156
- [Background] Denniff P, Spooner N. Volumetric absorptive microsampling: a dried sample collection technique for quantitative bioanalysis. Anal Chem. 2014 Aug 19;86(16):8489-95. doi: 10.1021/ac5022562. Epub 2014 Aug 6. PMID 25058158
- [Background] Roadcap B, Hussain A, Dreyer D, Carter K, Dube N, Xu Y, Anderson M, Berthier E, Vazvaei F, Bateman K, Woolf E. Clinical application of volumetric absorptive microsampling to the gefapixant development program. Bioanalysis. 2020 Jul;12(13):893-904. doi: 10.4155/bio-2020-0074. Epub 2020 Jul 10. PMID 32648772
- [Background] Fedoruk MN. Virtual drug testing: redefining sample collection in a global pandemic. Bioanalysis. 2020 Jun;12(11):715-718. doi: 10.4155/bio-2020-0119. Epub 2020 Jun 12. No abstract available. PMID 32530291
- [Background] Capiau S, Veenhof H, Koster RA, Bergqvist Y, Boettcher M, Halmingh O, Keevil BG, Koch BCP, Linden R, Pistos C, Stolk LM, Touw DJ, Stove CP, Alffenaar JC. Official International Association for Therapeutic Drug Monitoring and Clinical Toxicology Guideline: Development and Validation of Dried Blood Spot-Based Methods for Therapeutic Drug Monitoring. Ther Drug Monit. 2019 Aug;41(4):409-430. doi: 10.1097/FTD.0000000000000643. PMID 31268966
- [Background] Gaies E, Ben Sassi M, Charfi R, Salouage I, Jebabli N, ElJebari H, Klouz A, Daghfous R, Trabelsi S. Therapeutic durg monitoring of cyclosporin using area under the curve in nephrotic syndrome. Tunis Med. 2019 Feb;97(2):360-364. PMID 31539095
- [Background] Morales JM, Andres A, Rengel M, Rodicio JL. Influence of cyclosporin, tacrolimus and rapamycin on renal function and arterial hypertension after renal transplantation. Nephrol Dial Transplant. 2001;16 Suppl 1:121-4. doi: 10.1093/ndt/16.suppl_1.121. PMID 11369839
- [Background] Zhang X, Lin G, Tan L, Li J. Current progress of tacrolimus dosing in solid organ transplant recipients: Pharmacogenetic considerations. Biomed Pharmacother. 2018 Jun;102:107-114. doi: 10.1016/j.biopha.2018.03.054. Epub 2018 Mar 22. PMID 29550633
- [Background] Morales JM, Campistol JM, Kreis H, Mourad G, Eris J, Schena FP, Grinyo JM, Nanni G, Andres A, Castaing N, Brault Y, Burke JT. Sirolimus-based therapy with or without cyclosporine: long-term follow-up in renal transplant patients. Transplant Proc. 2005 Mar;37(2):693-6. doi: 10.1016/j.transproceed.2005.01.045. PMID 15848504
- [Background] Yoon HY, Hwang JJ, Kim DS, Song JW. Efficacy and safety of low-dose Sirolimus in Lymphangioleiomyomatosis. Orphanet J Rare Dis. 2018 Nov 14;13(1):204. doi: 10.1186/s13023-018-0946-8. PMID 30428897
- [Background] Mbughuni MM, Stevens MA, Langman LJ, Kudva YC, Sanchez W, Dean PG, Jannetto PJ. Volumetric Microsampling of Capillary Blood Spot vs Whole Blood Sampling for Therapeutic Drug Monitoring of Tacrolimus and Cyclosporin A: Accuracy and Patient Satisfaction. J Appl Lab Med. 2020 May 1;5(3):516-530. doi: 10.1093/jalm/jfaa005. PMID 32445361
- [Background] Kita K, Mano Y. Application of volumetric absorptive microsampling device for quantification of tacrolimus in human blood as a model drug of high blood cell partition. J Pharm Biomed Anal. 2017 Sep 5;143:168-175. doi: 10.1016/j.jpba.2017.05.050. Epub 2017 Jun 3. PMID 28601765
- [Background] Koster RA, Niemeijer P, Veenhof H, Hateren KV, Alffenaar JC, Touw DJ. A volumetric absorptive microsampling LC-MS/MS method for five immunosuppressants and their hematocrit effects. Bioanalysis. 2019 Mar;11(6):495-508. doi: 10.4155/bio-2018-0312. Epub 2019 Mar 20. PMID 30892068
- [Background] Paniagua-Gonzalez L, Diaz-Louzao C, Lendoiro E, Otero-Anton E, Cadarso-Suarez C, Lopez-Rivadulla M, Cruz A, de-Castro-Rios A. Volumetric Absorptive Microsampling (VAMS) for assaying immunosuppressants from venous whole blood by LC-MS/MS using a novel atmospheric pressure ionization probe (UniSpray). J Pharm Biomed Anal. 2020 Sep 10;189:113422. doi: 10.1016/j.jpba.2020.113422. Epub 2020 Jun 12. PMID 32590273
- [Background] Marshall DJ, Kim JJ, Brand S, Bryne C, Keevil BG. Assessment of tacrolimus and creatinine concentration collected using Mitra microsampling devices. Ann Clin Biochem. 2020 Sep;57(5):389-396. doi: 10.1177/0004563220948886. Epub 2020 Aug 20. PMID 32713180
- [Background] Scuderi C, Parker S, Jacks M, John GT, McWhinney B, Ungerer J, Mallett A, Healy H, Roberts J, Staatz C. Fingerprick Microsampling Methods Can Replace Venepuncture for Simultaneous Therapeutic Drug Monitoring of Tacrolimus, Mycophenolic Acid, and Prednisolone Concentrations in Adult Kidney Transplant Patients. Ther Drug Monit. 2023 Feb 1;45(1):69-78. doi: 10.1097/FTD.0000000000001024. PMID 36097333
- [Background] Freudenberger K, Hilbig U, Gauglitz G. Recent advances in therapeutic drug monitoring of immunosuppressive drugs. TrAC Trends Anal Chem. 2016;79:257-268. doi:10.1016/j.trac.2015.11.016